CLINICAL TRIAL: NCT05534698
Title: Coronary Artery Bypass Grafts or Percutaneous Coronary Intervention for Revascularization in Moderate to Highs Risk Patients With Ischemic Heart Disease and Reduced Left Ventricular Ejection Fraction
Brief Title: Coronary Artery Bypass Grafts or Percutaneous Coronary Intervention for High Risk Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-21000675
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: IHD; LV Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Intervention Model Description: Multicentre, open-label, parallel, randomized, controlled trial comparing revascularization by CABG versus by PCI in patients with severe CAD and at high risk
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI (Active Comparator): Revascularization by PCI
  Interventions: Procedure: PCI
- CABG (Active Comparator): Revascularization based on CABG.
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: PCI — Revascularization by PCI
  Arms: PCI
Procedure: CABG — Revascularization by CABG
  Arms: CABG

SUMMARY:
Most patients with Left Ventricular Systolic Dysfunction (LVSD) or heart failure (HF) have coronary artery disease (CAD) while some patients also have renal disease. Life-saving revascularization is underperformed in patients with LVSD or HF due to CAD, and especially if there is concomitant renal disease. We hypothesize that PCI will be non-inferior to CABG for all-cause mortality and recurrent myocardial infarction (MI), stroke or hospitalization for HF. To compare revascularization by PCI versus by CABG, we will perform a multicentre, open-label, parallel, randomized, controlled trial in patients with severe CAD who belong to defined categories of moderate-to-high risk characteristics, where guidelines acknowledge that both PCI and CABG are relevant treatment options.

DETAILED DESCRIPTION:
The STICH trial demonstrated a reduction in overall mortality after 10 years, but the 5-year analyses did not show significant benefits of CABG versus medical therapy. The extension of the STICH study, the STICHES study established the superiority of CABG over medical therapy for all-cause mortality (58.9% versus 66.1%; HR 0.84, 95%CI: 0.73-0.97; p = 0.02) over 9.8 years. Thus, these studies suggest that to offset the early operative risks of CABG, 10-year survival is needed. As many patients with HF and/or LVSD are elderly, both clinicians and patients are often unwilling to accept increased short-term risk even if they might eventually achieve long-term benefit, and thus not favour CABG. The available evidence suggest that PCI is feasible for patients with ischemic LVSD, and that PCI may yield long-term mortality rates like CABG with lower short-term morbidity The planned trial is a multicentre, open-label, parallel, randomized, controlled trial comparing revascularization by CABG versus by PCI in patients with severe CAD and at high risk, where guidelines accept both CABG and PCI as suitableand mortality. High risk is defined as patients with LVEF <45%, (irrespectively of clinical HF and severe renal disease), left anterior descending (LAD) disease in one- or two vessel disease, three-vessel disease with a SYNTAX score of up to 22 and left main disease with a SYNTAX score of up to 32.

The trial is powered for non-inferiorty.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

  * LVEF<45% with or without HF medication
  * Heart team believes that a meaningful revascularization can be achieve both by PCI and by CABG
  * Patients with severe CAD, where guidelines suggest equipoise between PCI and CABG

Exclusion Criteria:

* Decompensated HF requiring inotropic/adrenergic support, invasive or non-invasive ventilation or intra-aortic balloon pump/ ventricular assist device therapy less than 48 hours prior to randomization

  * Recent (< 1 month) ST-elevation myocardial infarction
  * Recent (< 1 month) type 2 myocardial infarction ▪ Valvular heart disease or any other cardiac conditions (for example, left ventricular aneurysm) indicating the need for surgical repair/replacement
  * Prohibitive bleeding risk or clinical scenario mandating avoidance of long-term dual antiplatelet therapy
  * Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1550 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality, stroke, MI and hospitalization for HF | up to 10 years with analysis after 5 years
  time to event

SECONDARY OUTCOMES:
Composite of occurrence of cardiovascular death or cardiovascular rehospitalization. | up to 10 years with analysis after 5 years
  time to event

OTHER OUTCOMES:
combined occurrence of major bleeding, new renal filtration and dialysis | up to 10 years with analysis after 5 years
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Lars V Køber, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data are available in a RedCap database and will be shared with other researchers after final report.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: up to 10 years
Access Criteria: For scientific purposes